CLINICAL TRIAL: NCT01859754
Title: Postmarketing Requirement Non-Interventional 2-armed Study to Evaluate the Safety of Octagam® Immune Globulin Intravenous (Human) 5% Liquid Preparation, With a Special Emphasis on Monitoring, Analysis and Reporting of Thromboembolic Events
Brief Title: Octagam 5% Versus Comparator Post Marketing Trial
Status: Completed | Type: Observational
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Other Study IDs: GAM5-28
Record Dates: First submitted 2013-05-09; First posted 2013-05-22 (Estimated); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Primary Immune Deficiency Disorder
Keywords: Primary Immune Deficiency Syndrome; Primary immunodeficiency Disease (PIDD); PID
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Octagam 5%: Primary Immune Deficiency Syndrome patients receiving Octagam 5% by infusion who have been treated with a marketed IVIG product for at least 6 months.
  Interventions: Biological: Octagam 5%
- Other marketed IVIG product: Primary Immune Deficiency Syndrome patients receiving marketed IVIG product other than Octagam 5% by infusion as treatment for at least 6 months.
  Interventions: Biological: Other marketed IVIG product

INTERVENTIONS:
Biological: Octagam 5% — Intravenous immunoglobulin 5%
  Groups: Octagam 5%
Biological: Other marketed IVIG product — Any intravenous immunoglobulin marketed product approved for the treatment of PID
  Groups: Other marketed IVIG product

SUMMARY:
Study Design:

This is a 2 arm non-interventional trial that will compare the occurrence of adverse drug reactions between Octagam 5% and other marketed IVIG infusion treatments.

DETAILED DESCRIPTION:
This Post Marketing Study is a prospective, 2-armed, multicenter, non-interventional study. Patients will either be administered the brand of IGIV therapy ordered by their prescribing physician, or for patients issued unspecified or generic prescriptions of IGIV therapy, octagam® 5% or another brand of IGIV therapy will be provided by the Investigator according to federal, state and local regulations and good clinical practice (GCP) guidelines.

The primary objective is to assess and evaluate the safety profile of octagam® 5% during or after administration under routine clinical use for all labeled indications, with a special emphasis on the occurrence of TEEs. The incidence of TEEs in patients receiving octagam® 5% will be compared with the incidence rate in a matching concurrent control group of patients receiving other IGIVs for routine clinical use.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18 years.
2. Patients with confirmed diagnosis of Primary Humoral Immunodeficiency (PI) as stated by the World Health Organization and requiring immunoglobulinreplacement therapy due to hypogammaglobulinemia or agammaglobulinemia.
3. Patients on regular treatment (every 3 to 4 weeks) with low dose IGIV (1 g/kg) for a period of at least 6 months without changing the brand.

Exclusion Criteria:

1. Patients with a history of TEEs within the previous 24 months.
2. Patients with a regular treatment frequency of more than once every 3 to 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old with Primary Immune Deficiency Syndrome PID receiving marketed IVIG as treatment
Sampling Method: Non-Probability Sample
Enrollment: 623 (Actual)
Dates: Start 2013-05-21 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
Incidence Rate of Thromboembolytic events | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Frenzel, Principal Investigator — International Medical Monitor, Octapharma AG
Locations (25):
- United States (25):
  - Octapharma Research Site, Granada Hills, California
  - Octapharma Research Site, Irvine, California
  - Octapharma Research Site, Los Angeles, California
  - Octapharma Research Site, Redlands, California
  - Octapharma Research Site, Centennial, Colorado
  - Octapharma Research Site, Roswell, Georgia
  - Octapharma Research Site, Chicago, Illinois
  - Octapharma Research Site, Springfield, Illinois
  - Octapharma Research Site, Fort Wayne, Indiana
  - Octapharma Research Site, Wichita, Kansas
  - Octapharma Research Site, Fort Mitchell, Kentucky
  - Octapharma Research Site, Farmington Hills, Michigan
  - Octapharma Research Site, Plymouth, Minnesota
  - Octapharma Research Site, Omaha, Nebraska
  - Octapharma Research Site, East Setauket, New York
  - Octapharma Research Site, New York, New York
  - Octapharma Research Site, Columbus, Ohio
  - Octapharma Research Site, Mayfield Heights, Ohio
  - Octapharma Research Site, Toledo, Ohio
  - Octapharma Research Site, Pawtucket, Rhode Island
  - Octapharma Research Site, Anderson, South Carolina
  - Octapharma Research Site, Nashville, Tennessee
  - Octapharma Research Site, Amarillo, Texas
  - Octapharma Research Site, Dallas, Texas
  - Octapharma Research Site, Irving, Texas